CLINICAL TRIAL: NCT05643989
Title: Randomized Non-inferiority Single-center Prospective Trial of Malignant Colonic Obstruction Therapy With Self-expandable Metal Stent (SEMS) Endoscopic Placement or Stoma Formation.
Brief Title: Self-expandable Metal Stent (SEMS) Endoscopic Placement for Malignant Colonic Obstruction Therapy
Acronym: PATENCY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34-20
Record Dates: First submitted 2022-06-10; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms,Colorectal
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-expandable metal stent (SEMS) endoscopic placement. (Active Comparator): Anesthesia will include only propofol injection. A covered or partially covered metal self- expanding stent is placed in the area of tumor stenosis by the conductor, symmetrically in relation to the area of tumor stenosis.
  Interventions: Procedure: Endoscopic self-expandable metal stent placement
- Stoma formation. (Placebo Comparator): Anesthetic care will include general endotracheal anesthesia with positioning of nasogastric tube and bladder catheterization. The diverting stoma formation will be proceed in 10 sm proximally to tumor.
  Interventions: Procedure: Stoma formation

INTERVENTIONS:
Procedure: Stoma formation — Trocar placement: the optical trocar (10 mm) will be inserted just near umbilicus . An abdominal revision is performed to determine the location of the tumor. Colon in 10 sm proximally to tumor is prepared for the discharge stoma formation. In the corresponding location on the anterior abdominal wall is formed incision of skin and subcutaneous tissue to the aponeurosis, the cut length is 2.5 sm. After that, aponeurosis crucial incision is performed. The previously prepared colon is brought out to the anterior abdominal wall with the help of a grasper. Discharge stoma is attached to a holding device; colon is fixed by the interrupted sutures (Polysorb 3-0). In the operating room, the stoma is opened, the intestinal patency is checked in both directions, and hemostasis is revealed. With the help of optics, the presence of intestinal tension is checked; if necessary, the colon is additionally mobilized.
  Arms: Stoma formation.
Procedure: Endoscopic self-expandable metal stent placement — The colonoscope is passed to the distal edge of the tumor and a biopsy of the tumor is performed (if the tumor has not previously been verified). Through the tumor stenosis radioscopically guided metal conductor with atraumatic distal end installs in the proximal colon. A covered or partially covered metal self- expanding stent is placed in the area of tumor stenosis by the conductor, symmetrically in relation to the area of tumor stenosis. Radioscopically and endoscopically guided disclosure of a SEMS is performed immediately after which there is an abundant discharge of gases and intestinal contents. Upon completion of the procedure, the patient is transferred to the patient's room. The next day, a control X-ray of the abdomen is taken.
  Arms: Self-expandable metal stent (SEMS) endoscopic placement.

SUMMARY:
Compare the effectiveness of Self-expandable metal stent (SEMS) and diverting stoma formation for the bowel preparation as a bridge to surgical treatment of patients with MCO.

DETAILED DESCRIPTION:
Surgical treatment of MCO is associated with high mortality and frequent development of postoperative complications. Stoma formation is the traditional method of urgent treatment of MCO. Currently there are more than 150 methods of colorectal stomas formation, but all of themare associated with a high risk of complications (10-20%), inclusively both early and late postoperative period. It results in longerhospital stay and requires additional financial expenses, also reoperations can be fatal for patients.

Analysis of recent publications devoted to the treatment of MCO shows increasing implemented of new strategies of patents management, such as "fast track surgery", or "fast track recovery strategy" in clinical practice. Minimally invasive endoscopic procedures as a first stage of MCO treatment leads to transformation of previously performed multi-stage surgical interventions into one - stage.

Development of up-to-date endoscopic science and technology provides a wide usage ofself-expandable metal stent (SEMS) in clinical practice. This strategy helps to avoid stoma formation or emergency surgery, becoming a "bridge" to a radical surgery.

There are currently no studies directly comparing discharge stoma with endoscopic self-expandable metal stenting in preparation for colorectal cancer radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are 18 years old or older
2. Stage I-IV according to TNM classification
3. Patients with malignant colonic obstruction
4. Overall health status according to ASA classification: I-III
5. Overall health status according to Charlson comorbidity index ≤ 8 points
6. Signed informed consent with agreement to attend all study visits
7. The patient is not pregnant

Exclusion Criteria:

1. Inflammatory bowel disease
2. Acute purulent process in the abdominal cavity
3. The patient wants to withdraw from the clinical trial
4. Loss to follow-up

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-05-11 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation (absence of feaces) according to Boston Bowel Preparation Scale | on the 3rd day after obstruction treatment (SEMS or stoma formation)
  Evaluated via colonoscopy in colon and rectum distal to the tumour. Total score of bowel preparation measured from 0 to 9. The maximum BBPS score for a perfectly clean colon without any residual liquid is 9 and the minimum BBPS score for an unprepared colon is 0. This is evaluated by the endoscopist

SECONDARY OUTCOMES:
Intraoperative complications rate during stoma formation or stent placement | 1 day (the day of procedure)
  The rate of complications during the procedure
Early postoperative complications rate after stoma formation or stent placement | up to 7 days after procedure
  The rate of complications after the procedure
Length of hospital stay after stoma formation or stent placement | 30 days after procedure
  Number of days spent in hospital after procedure
Quality of life before and after stoma formation or stent placement | -1 day (before procedure), 3rd and 7th day after procedure
  Measured by patient-reported SF-36 scale before and after procedure
Operation time of resectional surgery | 1 day (the day of tumor resection surgery )
  The duration of surgical procedure in minutes
Stoma formation rate | 1 day (the day of tumor resection surgery )
  The percentage of patients who had preventive or definitive stoma during resectional surgery in the SEMS group
Stoma reversal rate | 1 day (the day of tumor resection surgery )
  The rate of previously formed stoma reversal simultaneously with tumor resection
Early postoperative complications rate after resectional surgery | 30 days after resectional surgery
  The rate complications after tumor resection surgery
Length of hospital stay after resectional surgery | 30 days after resectional surgery
  Number of days spent in hospital after tumor resection surgery
Intraoperative complications rate during resectional surgery | 1 day (the day of resectional surgery)
  The rate of complications during tumor resection surgery
Late complications rate during resectional surgery | 31-90 days after tumor resection surgery
  The rate of complications after tumor resection surgery

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of colorectal and minimally invasive surgery University Hospital n2, Clinical Center Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronin KA, Lake AJ, Scott S, Sherman RL, Noone AM, Howlader N, Henley SJ, Anderson RN, Firth AU, Ma J, Kohler BA, Jemal A. Annual Report to the Nation on the Status of Cancer, part I: National cancer statistics. Cancer. 2018 Jul 1;124(13):2785-2800. doi: 10.1002/cncr.31551. Epub 2018 May 22. PMID 29786848
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Cheynel N, Cortet M, Lepage C, Benoit L, Faivre J, Bouvier AM. Trends in frequency and management of obstructing colorectal cancers in a well-defined population. Dis Colon Rectum. 2007 Oct;50(10):1568-75. doi: 10.1007/s10350-007-9007-4. PMID 17687610
- [Background] Baron TH. Colonic stenting: a palliative measure only or a bridge to surgery? Endoscopy. 2010 Feb;42(2):163-8. doi: 10.1055/s-0029-1243881. Epub 2010 Feb 5. PMID 20140833
- [Background] Larkin JO, Moriarity AR, Cooke F, McCormick PH, Mehigan BJ. Self-expanding metal stent insertion by colorectal surgeons in the management of obstructing colorectal cancers: a 6-year experience. Tech Coloproctol. 2014 May;18(5):453-8. doi: 10.1007/s10151-013-1073-0. Epub 2013 Oct 10. PMID 24114608
- [Background] Kim EJ, Kim YJ. Stents for colorectal obstruction: Past, present, and future. World J Gastroenterol. 2016 Jan 14;22(2):842-52. doi: 10.3748/wjg.v22.i2.842. PMID 26811630
- [Background] Maleckis K, Anttila E, Aylward P, Poulson W, Desyatova A, MacTaggart J, Kamenskiy A. Nitinol Stents in the Femoropopliteal Artery: A Mechanical Perspective on Material, Design, and Performance. Ann Biomed Eng. 2018 May;46(5):684-704. doi: 10.1007/s10439-018-1990-1. Epub 2018 Feb 22. PMID 29470746
- [Background] Nakata K, Fukunaga M, Ebihara T, Kato F, Amano K, Babaya A, Matsushita A, Furukawa H, Matsushima Y, Matsumoto H, Fujihara S, Kawabata R, Usui A, Yamamoto T, Oda K, Kawase T, Kimura Y, Nakata Y, Ohzato H. [A study of laparoscopic stoma creation for patients with malignant bowel obstruction]. Gan To Kagaku Ryoho. 2013 Nov;40(12):1702-4. Japanese. PMID 24393894
- [Background] van den Berg MW, Ledeboer M, Dijkgraaf MG, Fockens P, ter Borg F, van Hooft JE. Long-term results of palliative stent placement for acute malignant colonic obstruction. Surg Endosc. 2015 Jun;29(6):1580-5. doi: 10.1007/s00464-014-3845-7. Epub 2014 Oct 8. PMID 25294532
- [Result] Kim YW, Kim IY. The Role of Surgery for Asymptomatic Primary Tumors in Unresectable Stage IV Colorectal Cancer. Ann Coloproctol. 2013 Apr;29(2):44-54. doi: 10.3393/ac.2013.29.2.44. Epub 2013 Apr 30. PMID 23700570